CLINICAL TRIAL: NCT01327326
Title: Opioid Modulation of Two Models of Pain Inhibition in Healthy Controls and Patients With Temporomandibular Disorder (TMD)
Brief Title: Role of the Endogenous Opioid System Underlying Modulation of Experimental Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: American Pain Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: APS2011
Record Dates: First submitted 2011-03-24; First posted 2011-04-01 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Temporomandibular Disorder; Facial Pain
Keywords: Pain modulation; Experimental pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain | interventions — Naltrexone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMD patients (Active Comparator): Intervention:
  * Drug: Naltrexone
  * Drug: placebo
  Interventions: Drug: Naltrexone; Drug: Placebo
- Healthy controls (Active Comparator): Intervention:
  * Drug: Naltrexone
  * Drug: placebo
  Interventions: Drug: Naltrexone; Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — Oral, 50 mg, 1 Time Dose
  Other Names: Revia
Drug: Placebo — Oral, 1 Time Dose
  Other Names: Placebo/sugar pill

SUMMARY:
The aim of this proposal is to characterize pain inhibition in healthy controls and Temporomandibular Disorder (TMD) patients with two models of endogenous pain modulation (off-set analgesia; conditioned pain modulation), and to investigate the function of the endogenous opioid system in these responses by using pharmacological blockade of the opioid receptor.

DETAILED DESCRIPTION:
Dysfunction in endogenous pain inhibitory systems has been proposed as a factor in the development and maintenance clinical pain disorders particularly in Temporomandibular Disorder (TMD). Dysfunction has been observed with a model known as diffuse noxious inhibitory controls (DNIC), but other models that engage inhibitory systems (offset analgesia) have not been fully evaluated in chronic pain patients.

DNIC evaluates an individual's capacity to engage endogenous pain inhibition. The paradigm is a spatial inhibition model based on the principle that "pain-inhibits-pain" in which pain in a local area is inhibited by a second pain that can be anywhere else in the body. DNIC is traditionally studied by observing a reduction of pain produced by a focal pain stimulus (contact heat) as a result of a second painful stimulus. Research from our lab and others suggests that pain inhibition is reduced in a number of chronic pain conditions. The investigators preliminary data suggests that pain inhibition during DNIC is modulated in part by endogenous opioids; however, results from other DNIC studies have been mixed. In addition, it is possible that reductions in the ability to engage endogenous inhibitory systems in chronic pain patients are due to a weakening of the endogenous opioid system. While pharmacological studies have been conducted with healthy cohorts, only one study has examined the opioid involvement in chronic pain patients.

Offset analgesia is thought to reflect a form of temporal pain inhibition which is usually defined by three stimulus temperature phases: a baseline phase followed by a manipulation phase in which the temperature is briefly increased and returns to the baseline temperature during an "offset" phase. A reduction in pain ratings is observed approximately 15s after the temperature drop (third phase), which is ~50% lower than ratings at the same time point for "constant" trials that continued 48°C for 40s. No studies have examined offset analgesia in a chronic pain cohort or its sensitivity of opioid blockade.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-50 years old
* Controls: pain-free based on Research Diagnostic Criteria (RDC) exam
* TMD: chronic musculoskeletal pain (face) based on Research Diagnostic Criteria (RDC) exam

Exclusion Criteria:

* Inability to adequately communicate and understand informed consent form;
* Inability to reliably rate pain intensity;
* Uncontrolled hypertension (or receiving treatment for hypertension with BP of greater than 140/95);
* Serious systemic (e.g. Diabetes, thyroid problems, etc.);
* Serious cardiovascular/pulmonary disease;
* Neurological problems with significant changes in somatosensory and pain perception at the intended stimulation sites (hand, foot);
* Serious psychiatric problems requiring treatment (schizophrenia, bipolar disorder);
* Other chronic pain conditions (e.g., low back pain, fibromyalgia);
* Any other ongoing acute pain problem (arthritis, injury-related pain); or,
* Irregular menstrual cycles (>40 days) or menstrual cycle disorders (e.g. PMS, dysmenorrhea).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Post-drug efficacy of pain inhibition | 1 hour after study medication (day 1)
  A change in the ability to reduce experimental pain sensitivity during two models of pain inhibition will be evaluated before and after medication.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D King, PhD, Principal Investigator — University of Florida